CLINICAL TRIAL: NCT01013662
Title: Tight Glycemic Control and Sepsis Related Dyslipidemia
Brief Title: Lipid Profile in Patients With Severe Sepsis or Septic Shock Under Strict or Liberal Glycemic Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Francisco Garcia Soriano, Universidade de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: scap1501
Record Dates: First submitted 2009-11-13; First posted 2009-11-16 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2009-11

CONDITIONS: Septic Shock; Sepsis
Keywords: septic shock; glycemic control; icu; lipid metabolism; septic patients
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Glycemic Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- glycemic control between 180 and 220 mg/dl (Active Comparator)
  Interventions: Procedure: glycemic control
- glycemic control for levels between 80 and 110 mg/dl (Active Comparator)
  Interventions: Procedure: glycemic control

INTERVENTIONS:
Procedure: glycemic control — exogenous insulin

SUMMARY:
Study of the lipid metabolism under glycemic control in septic patients who got an university 14 bed ICU.

Hypothesis: establish a relationship between lipid metabolism alterations and glycemic control or infusion of exogenous insulin

DETAILED DESCRIPTION:
The investigators enrolled 69 consecutive patients with severe sepsis or septic shock and divided them in two different groups after randomization with sealed envelopes.

One group called intensive glycemic control with glycemic levels been between 80 to 110 mg/dl with exogenous insulin.

The other group called conventional glycemic control with glycemic levels been between 180 and 220 mg/dl.

Blood samples were collected at 0, 12, 24, 48 and 72 hours to measure HDL, LDL, Total cholesterol, free fatty acids and oxidized LDL.

Clinical data as creatinine, P/F ratio, bilirubins, platelets, lactate, arterial blood gasometry were either monitored.

ELIGIBILITY:
Inclusion Criteria:

* all patients aged between 18 and 80 years old
* with the diagnostic of septic shock or severe sepsis

Exclusion Criteria:

* pregnants,
* previous diagnosis of any cancer,
* diagnosis of leptospirosis,
* diagnosis of aids.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2005-01; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
establish a relationship between lipid metabolism alterations and glycemic control | 2 years

REFERENCES:
- [Derived] Cappi SB, Noritomi DT, Velasco IT, Curi R, Loureiro TC, Soriano FG. Dyslipidemia: a prospective controlled randomized trial of intensive glycemic control in sepsis. Intensive Care Med. 2012 Apr;38(4):634-41. doi: 10.1007/s00134-011-2458-z. Epub 2012 Feb 2. PMID 22297666